CLINICAL TRIAL: NCT04694326
Title: The Incidence of Diabetes Unawareness in Patients Hospitalized Outside Internal Medicine Services and Related Factors: A Multidisciplinary Study for Detecting Undiagnosed Diabetes
Brief Title: The Incidence of Diabetes Unawareness in Patients Hospitalized Outside Internal Medicine Services and Related Factors
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: INPATİENTA1C
Record Dates: First submitted 2021-01-01; First posted 2021-01-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-01

CONDITIONS: Diabetes; Hba1c; Inpatient Facililty Diagnoses
Keywords: Diabetes Mellitus; Diabetes Unawareness; İnpatient; HbA1c
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inpatients: Patients who were inpatients of units other than internal medicine services and internal medicine side-branch services
  Interventions: Diagnostic Test: HbA1c

INTERVENTIONS:
Diagnostic Test: HbA1c — The participants' age, sex, education level, known diseases, unit of hospitalization and inpatient diagnosis were questioned and recorded. Height, weight and waist circumference measurements were taken. Fasting blood sugar and HbA1c measurements were made
  Other Names: Anthropometric measures; Glucose

SUMMARY:
Our purpose is to determine the prevalence of undiagnosed diabetes by checking HbA1c in patients hospitalized outside internal medicine services and assess whether or not there is a difference between those without diabetes awareness and those with known diabetes in terms of age, sex, education status, presence of comorbidity and Body Mass Index (BMI).

DETAILED DESCRIPTION:
The study included 630 patients hospitalized outside internal medicine services and internal medicine side-branch services at or over the age of 18 whose anthropometric measurements could be made. The sociodemographic properties and comorbidities of the patients were recorded. Their anthropometric measurements, fasting blood glucose and HbA1c measurements were made. Those with a previous diagnosis of diabetes were grouped as 'Known Diabetes', those without a known diabetes diagnosis but with an HbA1c value of ≥6.5% during hospitalization were grouped as 'Diabetes Unaware', and those with an HbA1C value of <6.5% were grouped as 'No Diabetes'. Whether or not there were differences among the 3 groups based on sociodemographic characteristics, anthropometric measurements and disease statuses was examined.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients of units other than internal medicine services and internal medicine side-branch services at or
* Over the age of 18
* Anthropometric measurements could be made were included

Exclusion Criteria:

* Had comorbidities that could affect their anthropometric measurements (heart failure, edema, liver cirrhosis, cancer, cachexia, Cushing syndrome, etc.),
* Who had been using steroids for more than a month,
* Pregnant
* Postoperative period

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study was conducted at two different tertiary healthcare institutions located in Istanbul in Turkey. Patientswho were inpatients of units other than internal medicine services and internal medicine side-branch services at or over the age of 18 whose anthropometric measurements could be made were included. . The internal units included neurology, dermatology, physiotherapy and rehabilitation, cardiology, infectious diseases and pulmonology services, while the surgical units included general surgery, cardiovascular surgery, pulmonary surgery, orthopedics and traumatology, brain surgery, ophthalmology, urology, gynecology and plastic surgery services.
Sampling Method: Non-Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Diabetes Unawaraness Prevalance | 14 days
  Diabetes unawaraness prevalance in inpatient settings

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Abdülhamid Han Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No